CLINICAL TRIAL: NCT04305457
Title: Nitric Oxide Gas Inhalation Therapy in Spontaneous Breathing Patients With Mild/Moderate COVID-19: a Randomized Clinical Trial
Brief Title: Nitric Oxide Gas Inhalation Therapy for Mild/Moderate COVID-19
Acronym: NoCovid
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: COVID wave passed
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Lorenzo Berra, MD, Medical Doctor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NOgas mildCOVID-19
Record Dates: First submitted 2020-03-09; First posted 2020-03-12 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Coronavirus Infections; Pneumonia, Viral; Acute Respiratory Distress Syndrome
Keywords: COVID-19; ARDS; Mechanical Ventilation; Nitric Oxide
MeSH Terms: conditions — Coronavirus Infections; Pneumonia, Viral; Respiratory Distress Syndrome; COVID-19 | interventions — Nitric Oxide

STUDY DESIGN:
Intervention Model Description: This study includes a randomized, parallel arm clinical trial in which subjects will be randomized to receive either inhaled nitric oxide (in addition to the standard of care) or the standard of care alone.
  In a third arm, COVID-19 subjects will be enrolled at Providence HealthCare Network, Anchorage (AK). Subjects in this arm will not be randomized and will all receive nitric oxide gas either as an inpatient or outpatient.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Nitric Oxide inhalation (Experimental): Nitric Oxide will be delivered through a non invasive CPAP system (with minimal pressure support to decrease discomfort due to the facial mask) or through a non-rebreathing mask system.
  Interventions: Drug: Nitric Oxide
- Control (No Intervention): Patients assigned to the control group will not receive any gas therapy.
- Nitric Oxide Inhalation (Non-Randomized) (Experimental): All subjects part of this arm will receive nitric oxide gas either as an inpatient or outpatient. Nitric Oxide will be delivered through a non invasive CPAP system (with minimal pressure support to decrease discomfort due to the facial mask) or through a non-rebreathing mask system. Patients in this arm will not be randomized, so that all patients receive the study medication.
  Interventions: Drug: Nitric Oxide

INTERVENTIONS:
Drug: Nitric Oxide — Nitric Oxide (NO) will be delivered together with the standard of care for a period of 20-30 minutes 2 times per day for 14 consecutive days from time of enrollment. Targeted No inhaled concentration will be maintained between 140 and 180 ppm. The gas will be delivered through a CPAP circuit ensuring an end-expiratory pressure between 2 and 10 cmH2O or through a non-rebreathing mask without positive end-expiratory pressure, depending on the clinical needs of the subject.
  Other Names: Nitric Oxide inhalation
  Arms: Nitric Oxide Inhalation (Non-Randomized); Nitric Oxide inhalation

SUMMARY:
The scientific community is in search for novel therapies that can help to face the ongoing epidemics of novel Coronavirus (SARS-Cov-2) originated in China in December 2019. At present, there are no proven interventions to prevent progression of the disease. Some preliminary data on SARS pneumonia suggest that inhaled Nitric Oxide (NO) could have beneficial effects on SARS-CoV-2 due to the genomic similarities between this two coronaviruses. In this study we will test whether inhaled NO therapy prevents progression in patients with mild to moderate COVID-19 disease.

DETAILED DESCRIPTION:
To date, no targeted therapeutic treatments for the ongoing COVID-19 outbreak have been identified. Antiviral combined with adjuvant therapies are currently under investigation. The clinical spectrum of the infection is wide, ranging from mild signs of upper respiratory tract infection to severe pneumonia and death.

In the patients who progress, the time period from symptoms onset to development of dyspnea is reported to be between 5 to 10 days, and that one to severe respiratory distress syndrome from 10 to 14 days. Globally, 15 to 18% of patients deteriorates to the need of mechanical ventilation, despite the use of non-invasive ventilatory support in the earliest phases of the disease. Probability of progression to end stage disease is unpredictable, with the majority of these patients dying from multi-organ failure. Preventing progression in spontaneously breathing patients with mild to moderate disease would translate in improved morbidity and mortality and in a lower use of limited healthcare resources.

In 2004, during the SARS-coronavirus (SARS-CoV) outbreak, a pilot study showed that low dose ( max 30 ppm) inhaled NO for 3 days was able to shorten the time of ventilatory support. At the same time, NO donor compound S-nitroso-N-acetylpenicillamine increased survival rate in an in-vitro model of SARS-CoV infected epithelial cells.Based on the genetic similarities between the two viruses, similar effects of NO on SARS-CoV-2 can be hypothesized. While further in-vitro testing is recommended, we proposed a randomized clinical trial to test the effectiveness of inhaled NO in preventing the progression of SARS-CoV-2 related disease, when administered at an early stage.

ELIGIBILITY:
Inclusion Criteria:

1. Laboratory confirmed COVID19 infection defined with a positive RT-PCR from any specimen and/or detection of SARS-CoV-2 IgM/IgG antibodies.
2. Hospital admission with at least one of the following:

   1. fever ≥ 36.6 °C from axillary site; or ≥ 37.2°C from oral site; or ≥ 37.6°C from tympanic or rectal site.
   2. Respiratory rate ≥ 24 bpm
   3. cough
3. Spontaneous breathing with or without hypoxia of any degree. Gas exchange and ventilation maybe assisted by any continuous continuous airway pressure (CPAP), or any system of Non Invasive Ventilation (NIV), with Positive End-Expiratory Pressure (PEEP) ≤ 10 cmH2O.

Exclusion Criteria:

1. Tracheostomy
2. Therapy with high flow nasal cannula
3. Any clinical contraindications, as judged by the attending physician
4. Patients enrolled in another interventional study
5. Hospitalized and confirmed diagnosis of COVID-19 for more than 72 hours
6. Previous intubation for COVID-19
7. Patient not committed to full support (DNR, DNI or CMO)
8. Patient requiring oxygen at home for lung comorbidities
9. Primary cause of hopitalization not due to COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-03-21 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
Reduction in the incidence of patients with mild/moderate COVID-19 requiring intubation and mechanical ventilation | 28 days
  The primary outcome will be the reduction in the incidence of patients requiring intubation and mechanical ventilation, as a marker of deterioration from a mild to a severe form of COVID-19. Patients with indication to intubation and mechanical ventilation but concomitant DNI (Do Not Intubate) or not intubated for any other reason external to the clinical judgment of the attending physician will be considered as meeting the criteria for the primary endpoint.

SECONDARY OUTCOMES:
Mortality | 28 days
  Proportion of deaths from all causes
Time to clinical recovery | 28 days
  Time from initiation of the study to discharge or to normalization of fever (defined as <36.6°C from axillary site, or < 37.2°C from oral site or < 37.8°C from rectal or tympanic site), respiratory rate (< 24 bpm while breathing room air), alleviation of cough (defined as mild or absent in a patient reported scale of severe >>moderate>>mild>>absent) and resolution of hypoxia (defined as SpO2 ≥ 93% in room air or P/F ≥ 300 mmHg). All these improvements must be sustained for 72 hours.

OTHER OUTCOMES:
Negative conversion of COVID-19 RT-PCR from upper respiratory tract | 7 days
  Proportion of patients with a negative conversion of RT-PCR from an oropharyngeal or oropharyngeal swab.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Berra, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Providence HealthCare Network, Anchorage, Alaska
  - Louisiana State University Health Shreveport, Shreveport, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts